CLINICAL TRIAL: NCT00073528
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase III Study Comparing GW572016 and Letrozole Versus Letrozole in Subjects With Estrogen/Progesterone Receptor- Positive Advanced or Metastatic Breast Cancer
Brief Title: Study Comparing Lapatinib (GW572016) And Letrozole Versus Letrozole In Subjects With Advanced Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGF30008; CLAP016A2308 (Other: Novartis); 2004-003928-35 (EudraCT Number); NCT00084968 (obsolete NCT alias)
Record Dates: First submitted 2003-11-24; First posted 2003-11-26 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasms
Keywords: Lapatinib; Letrozole; breast carcinoma; breast cancer; breast lump; HER2 positive metastatic breast cancer; breast cancer positive for human epidermal growth factor receptor 2; HER2; breast cancer progression; estrogen-receptor positive breast cancer; ER
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Letrozole 2.5 mg (Placebo Comparator): Letrozole (2.5 mg once daily orally) with Placebo (which matched with Lapatinib tablet)
  Interventions: Drug: Letrozole; Drug: Placebo
- Lapatinib 1500 mg + Letrozole 2.5 mg (Experimental): Lapatinib (1500 mg once daily orally) with Letrozole (2.5 mg once daily orally)
  Interventions: Drug: Lapatinib; Drug: Letrozole

INTERVENTIONS:
Drug: Lapatinib — 1500 mg orally once a day
  Other Names: GW572016
  Arms: Lapatinib 1500 mg + Letrozole 2.5 mg
Drug: Letrozole — 2.5 mg orally once a day
Drug: Placebo — Placebo (which matched with lapatinib tablet)
  Arms: Placebo + Letrozole 2.5 mg

SUMMARY:
This study evaluated and compared the efficacy and tolerability of lapatinib and letrozole, with letrozole and placebo in post-menopausal women with hormone receptor positive (ER positive and/or PgR positive) advanced or metastatic breast cancer, who had not received prior therapy for advanced or metastatic disease.

DETAILED DESCRIPTION:
Subjects were randomly assigned to receive either lapatinib (1500 mg once daily orally) with letrozole (2.5 mg once daily orally), or letrozole (2.5 mg once daily orally) with placebo (which matched with lapatinib tablet). Randomization was stratified by site of disease (i.e., soft tissue/visceral disease versus bone only disease) and time since prior adjuvant endocrine therapy (<6 months or ≥ 6 months from discontinuation of adjuvant anti-estrogen therapy (e.g. tamoxifen or raloxifene) or no prior adjuvant antiestrogen therapy). Study therapy was administered daily until disease progression (objective or symptomatic) or withdrawal from therapy (e.g., due to unacceptable toxicity, withdrawal of consent, or other reason). All subjects were to be followed for survival information until death.

On 13 Apr 2015, after the introduction of the Long Term Follow UP (LTFU) phase (per protocol amendment 07), subjects receiving study treatment with lapatinib plus letrozole, or letrozole plus placebo had continued access to this study treatment until the occurrence of one of the following criteria:

* Disease progression (as determined by the Investigator),
* Intercurrent illness that prevented further administration of study treatment
* Drug related AE which was considered by the investigator to warrant permanent discontinuation of study treatment
* The subject decided to withdraw from the study. Investigators collected AEs and/or SAEs related to study participation, until 30 days following study treatment discontinuation. Subjects who were being followed-up for OS but were not taking study medication, were withdrawn from the study.

The study was terminated on 22-Mar-2018 (last subject last visit).

ELIGIBILITY:
Key inclusion criteria

1. Signed informed consent;
2. Subjects with histologically confirmed invasive breast cancer with stage IV disease at primary diagnosis or at relapse after curative-intent surgery;

   * Subjects with either measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST).
   * If the disease was restricted to a solitary lesion, its neoplastic nature was confirmed by cytology or histology.
3. Tumors that were ER+ and/or PgR+;
4. Post-menopausal female subjects ≥ 18 years of age.
5. ECOG Performance Status of 0 or 1;
6. Subjects who had archived tumor tissue available to compare tumor response with intra-tumoral expression of ErbB1 and ErbB2.
7. Adjuvant therapy with an aromatase inhibitor and / or trastuzumab was allowed; however, treatment was to stop more than 1 year prior (>12 months) to the first dose of randomized therapy.
8. Subjects must have ended hormonal replacement therapy (HRT) at least 1 month (30 days) prior to receiving the first dose of randomized therapy.

Key exclusion criteria:

1. Pre-menopausal, pregnant, or lactating;
2. Received prior chemotherapy, hormonal therapy, immunotherapy, biologic therapy, or anti-ErbB1/ErbB2 therapy for advanced or metastatic disease;
3. Bisphosphonate therapy for bone metastases was allowed; however, treatment was to be initiated prior to the first dose of randomized therapy. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, was not permitted;
4. Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of randomized therapy (lapatinib or placebo);
5. Subjects with known history of/clinical evidence of CNS metastases or leptomeningeal carcinomatosis; and / or subjects on concurrent anti-cancer therapies other than letrozole; and / or who have not recovered from toxicities related to prior adjuvant therapy (surgery, radiotherapy, chemotherapy etc.)
6. Subjects with active or uncontrolled infection and/ or with history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1286 (Actual)
Dates: Start 2003-12-09 (Actual); Primary Completion 2008-06-03 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (237):
- United States (81):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Alhambra, California
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Montebello, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Oxnard, California
  - Novartis Investigative Site, Pleasant Hill, California
  - Novartis Investigative Site, Porterville, California
  - Novartis Investigative Site, Redondo Beach, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Santa Maria, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Vista, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Longmont, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Lakeland, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Port Saint Lucie, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Bettendorf, Iowa
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Robbinsdale, Minnesota
  - Novartis Investigative Site, Saint Louis Park, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Santa Fe, New Mexico
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, West Columbia, South Carolina
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Irving, Texas
  - Novartis Investigative Site, Ogden, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Charleston, West Virginia
- Argentina (2):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (5):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Douglas, Queensland
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Redcliffe, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
- Brazil (2):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (9):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Novartis Investigative Site, Santiago, Región Metro de Santiago, Chile
- Novartis Investigative Site, Bogotá, Colombia
- Croatia (3):
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Pula
  - Novartis Investigative Site, Split
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Prague
- Denmark (7):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Hillerød
  - Novartis Investigative Site, Koebenhavn Oe
  - Novartis Investigative Site, Næstved
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Vejle
- France (9):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse Cedex9
  - Novartis Investigative Site, Villejuif
- Germany (33):
  - Novartis Investigative Site, Aalen, Baden-Wurttemberg
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Heidenheim, Baden-Wurttemberg
  - Novartis Investigative Site, Schwetzingen, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Rehling, Bavaria
  - Novartis Investigative Site, Rosenheim, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Leer, Lower Saxony
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Coesfeld, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Ibbenbueren, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Altenkirchen, Rhineland-Palatinate
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Pinneberg, Schleswig-Holstein
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Tatabánya
- Ireland (6):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dooradoyle
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, Tallaght, Dublin
  - Novartis Investigative Site, Wilton, Cork
- Italy (6):
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Parma, Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Crema, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
- Mexico (4):
  - Novartis Investigative Site, Acapulco de Juárez, Guerrero
  - Novartis Investigative Site, Colima
  - Novartis Investigative Site, Durango
  - Novartis Investigative Site, Mexico City
- Netherlands (11):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Doetinchem
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Leidschendam
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Sittard-geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Christchurch, New Zealand
- Pakistan (2):
  - Novartis Investigative Site, Lahore
  - Novartis Investigative Site, Rawalpindi
- Peru (2):
  - Novartis Investigative Site, Callao
  - Novartis Investigative Site, Lima
- Poland (5):
  - Novartis Investigative Site, Bydogoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Africa (4):
  - Novartis Investigative Site, Capital Park
  - Novartis Investigative Site, Panorama
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Port Elizabeth
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seodaemun-gu, Seoul
  - Novartis Investigative Site, Seoul
- Spain (15):
  - Novartis Investigative Site, Alcala de Henares (Madrid)
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Elche
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Leganes, Madrid
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Móstoles
  - Novartis Investigative Site, Oviedo
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Vigo ( Pontevedra)
  - Novartis Investigative Site, Zaragoza
- Tunisia (3):
  - Novartis Investigative Site, Sfax
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (8):
  - Novartis Investigative Site, Chelmsford, Essex
  - Novartis Investigative Site, Manchester, Lancashire
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Huddersfield
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Johnston S, Pippen J Jr, Pivot X, Lichinitser M, Sadeghi S, Dieras V, Gomez HL, Romieu G, Manikhas A, Kennedy MJ, Press MF, Maltzman J, Florance A, O'Rourke L, Oliva C, Stein S, Pegram M. Lapatinib combined with letrozole versus letrozole and placebo as first-line therapy for postmenopausal hormone receptor-positive metastatic breast cancer. J Clin Oncol. 2009 Nov 20;27(33):5538-46. doi: 10.1200/JCO.2009.23.3734. Epub 2009 Sep 28. PMID 19786658
- [Background] Schwartzberg LS, Franco SX, Florance A, O'Rourke L, Maltzman J, Johnston S. Lapatinib plus letrozole as first-line therapy for HER-2+ hormone receptor-positive metastatic breast cancer. Oncologist. 2010;15(2):122-9. doi: 10.1634/theoncologist.2009-0240. Epub 2010 Feb 15. PMID 20156908
- [Background] Sherrill B, Amonkar MM, Sherif B, Maltzman J, O'Rourke L, Johnston S. Quality of life in hormone receptor-positive HER-2+ metastatic breast cancer patients during treatment with letrozole alone or in combination with lapatinib. Oncologist. 2010;15(9):944-53. doi: 10.1634/theoncologist.2010-0012. Epub 2010 Aug 26. PMID 20798196
- [Background] Finn RS, Press MF, Dering J, O'Rourke L, Florance A, Ellis C, Martin AM, Johnston S. Quantitative ER and PgR assessment as predictors of benefit from lapatinib in postmenopausal women with hormone receptor-positive, HER2-negative metastatic breast cancer. Clin Cancer Res. 2014 Feb 1;20(3):736-43. doi: 10.1158/1078-0432.CCR-13-1260. Epub 2013 Nov 6. PMID 24198242
- [Background] Prat A, Cheang MC, Galvan P, Nuciforo P, Pare L, Adamo B, Munoz M, Viladot M, Press MF, Gagnon R, Ellis C, Johnston S. Prognostic Value of Intrinsic Subtypes in Hormone Receptor-Positive Metastatic Breast Cancer Treated With Letrozole With or Without Lapatinib. JAMA Oncol. 2016 Oct 1;2(10):1287-1294. doi: 10.1001/jamaoncol.2016.0922. PMID 27281556
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 212 centers in 29 countries (Argentina, Australia, Brazil, Bulgaria, Canada, Chile, Colombia, Croatia, Czech Republic, Denmark, France, Germany, Hungary, Ireland, Italy, Republic of Korea, Mexico, Netherlands, New Zealand, Pakistan, Peru, Poland, Russian Federation, South-Africa, Spain, Tunisia, Turkey, UK, USA).
Groups:
- Placebo + Letrozole 2.5 mg: Participants received 6 tablets of placebo, identical in appearance to lapatinib tablets, orally daily (approximately at the same time each day), either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received 1 tablet of letrozole 2.5 milligrams (mg) orally daily, preferably with the daily dose of lapatinib.
- Lapatinib 1500 mg + Letrozole 2.5 mg: Participants received 6 tablets of Lapatinib orally daily (250 mg lapatinib/tablet for a total of 1500 mg of lapatinib/day; approximately at the same time each day), either 1 hour (or more) before breakfast or 1 hour (or more) after breakfast. Participants also received 1 tablet of letrozole 2.5 mg orally daily, preferably with the daily dose of lapatinib.
Period: Overall Study
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Started (All participants included in the Intent-To-Treat (ITT) population) | 644 | 642
Completed | 14 | 14
Not Completed | 630 | 628
Not completed — Death | 488 | 473
Not completed — Lost to Follow-up | 52 | 45
Not completed — Withdrawal by Subject | 50 | 45
Not completed — Study terminated by Sponsor | 10 | 29
Not completed — Other | 18 | 19
Not completed — Other | 9 | 12
Not completed — Protocol Violation | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg | Total
Number analyzed (Participants) | 644 | 642 | 1286
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.95) | 62.8 (9.70) | 63.1 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 644 | 642 | 1286
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 557 | 529 | 1086
  Black | 10 | 17 | 27
  Asian | 30 | 30 | 60
  American Hispanic | 44 | 57 | 101
  Other | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS) in the Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced or Metastatic Breast Cancer as Assessed by the Investigator
Description: PFS is defined as the time from randomization until the earliest date of disease progression (PD) or death due to any cause, if sooner. The date of documented PD is defined as the date of radiological PD as assessed by the investigator based on imaging data and also by the clinical assessment of symptomatic progression. Per Response Evaluation Criteria in Solid Tumors (RECIST 1.0), PD is defined as a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as a reference the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until the date of the first documented progression or date of death from any cause, whichever came first, assessed for up to 46 months
Population: HER2-Positive Population: all randomized participants who had documented amplification of baseline HER2 by fluorescence in situ hybridization (FISH) (=>2.0) or 3+ immunohistochemistry (IHC) (or 2+ IHC and FISH +) in archived tumor tissue regardless of whether or not study treatment had been received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Participants | 89 | 88
Statistical Analysis 1: Comparison: Placebo + Letrozole 2.5 mg vs Lapatinib 1500 mg + Letrozole 2.5 mg; Test type: Superiority or Other; p = 0.019, Log Rank — p-value is from stratified log-rank test, stratifying for site of disease and time since prior adjuvant endocrine therapy at screening; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.53 to 0.96] — The estimate of the treatment Hazard Ratio wase based on the log-rank test

2. Primary Outcome: Progression Free Survival (PFS) of Participants in the HER2-Positive Population as Assessed by the Investigator
Description: PFS is defined as the time from randomization until the earliest date of disease progression or death due to any cause, if sooner. The date of documented disease progression is defined as the date of radiological disease progression as assessed by the investigator based on imaging data and also by the clinical assessment of symptomatic progression. Per RECIST 1.0, disease progression is defined as a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 46 months
Population: HER2-Positive Population. Only those participants who experienced disease progression or died during their participation in the study were assessed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 89 | 88
Weeks | 13.0 [12.0 to 23.7] | 35.4 [24.1 to 39.4]
Statistical Analysis 1: Comparison: Placebo + Letrozole 2.5 mg vs Lapatinib 1500 mg + Letrozole 2.5 mg; Test type: Superiority or Other; p = 0.019, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.53 to 0.96] — The estimate of the treatment Hazard Ratio was based on the log-rank test

3. Secondary Outcome: Number of Participants With PFS in the Intent-To-Treat (ITT) Population as Assessed by the Investigator
Description: as for outcome 2
Time Frame: as for outcome 2
Population: ITT Population: all randomized participants, regardless of whether or not study treatment had been received. The ITT Population included the HER2-Positive Population, the HER2-Negative Population, and the HER2-Missing Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants | 476 | 413

4. Secondary Outcome: PFS in Participants in the ITT Population as Assessed by the Investigator
Description: as for outcome 2
Time Frame: as for outcome 2
Population: ITT Population. Only those participants who experienced disease progression or died during their participation in the study were assessed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 476 | 413
Weeks | 47.0 [36.9 to 50.9] | 51.7 [47.6 to 59.6]

5. Secondary Outcome: Overall Survival in the HER2-Positive Population
Description: Overall survival was defined as the time from randomization until death due to any cause.
Time Frame: From date of randomization until date of death due to any cause, assessed up to 46 months
Population: HER2-Positive Population. Only those participants who died during the study due to any cause were assessed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Weeks | 140.3 [92.1 to 159.4] | 144.7 [95.6 to NA] — NA: Not estimable due to insufficient number of participants with events

6. Secondary Outcome: Overall Tumor Response (OR) for Participants With Measurable and Non-measurable Disease, Including Bone Scans, in the HER2-Positive Population as Assessed by the Investigator
Description: OR is defined as the percentage of participants achieving either a confirmed complete response (CR) or partial response (PR). Response was assessed via Response Evaluation criteria in Solid Tumors (RECIST). The percentage of participants with response was calculated by using the formula: 100 * (number of participants with CR + number of participants with PR)/total number of participants. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the baseline sum LD.
Time Frame: Up to 46 months
Population: HER2-Positive Population
Measure: Number (95% Confidence Interval); unit: Percent response rate
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Percent response rate | 14.8 [8.7 to 22.9] | 27.9 [19.8 to 37.2]

7. Secondary Outcome: Number of Participants With Overall Tumor Response (OR) by Stratification Factors With Measurable Disease, Including Bone Scans, in the HER2-Positive Population as Assessed by the Investigator
Description: Participants were stratified based on site of disease at screening (SDS) (soft tissue or visceral or bone-only disease) and prior adjuvant endocrine therapy (PAET) (discontinuation interval [DI] =>6 months or DI <6 months). OR is defined as the number of participants achieving either a confirmed CR or PR. Response was assessed via RECIST. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the baseline sum LD. DI is defined as the time period from stopping the PEAT to the randomization date.
Time Frame: Up to 46 months
Population: HER2-Positive Population. Only those participants with measurable disease, including bone scans, were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 75 | 93
Participants
  SDS, Soft tissue or visceral | 14 | 31
  SDS, Bone-only disease | 0 | 0
  PAET, DI =>6 months: number analyzed (Participants) | 53 | 61
  PAET, DI =>6 months | 12 | 24
  PAET, DI <6 months: number analyzed (Participants) | 22 | 32
  PAET, DI <6 months | 2 | 7

8. Secondary Outcome: Clinical Benefit (CB) in the HER2-Positive Population as Assessed by the Investigator
Description: CB is defined as the percentage of participants with evidence of confirmed CR, PR, or stable disease (SD) for at least 6 months. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the baseline sum LD. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the baseline measurement.
Time Frame: Up to 46 months
Population: HER2-Positive Population
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Months | 28.7 [20.4 to 38.2] | 47.7 [38.2 to 57.4]

9. Secondary Outcome: Number of Participants With the Indicated Best Response From the Participants With Measurable and Non-measurable Disease, Including Bone Scans, in the HER2-Positive Population as Assessed by the Investigator.
Description: CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference the smallest sum LD since the baseline measurement. The best overall response is defined as the best response recorded from the start of treatment until disease progression/recurrence. PD: presence of target lesions, non-target lesions, and/or new lesions.
Time Frame: Up to 46 months
Population: HER2-Positive Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Participants
  CR | 4 | 5
  PR | 12 | 26
  SD | 35 | 44
  PD | 49 | 30
  Unknown | 8 | 6

10. Secondary Outcome: Number of Participants With the Indicated Best Response From the Participants With Measurable and Non-measurable Disease, Including Bone Scans, in the ITT Population as Assessed by the Investigator.
Description: as for outcome 9
Time Frame: Up to 46 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants
  CR | 26 | 28
  PR | 153 | 168
  SD | 243 | 280
  PD | 174 | 113
  Unknown | 48 | 53

11. Secondary Outcome: Number of Participants With the Indicated Time to Response for CR or PR in the HER2-Positive Population as Assessed by the Investigator
Description: Time to response is defined as the time from randomization until the first documented evidence of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sume of the LD of target lesions, taking as reference the baseline sum LD) (whichever status was recorded first). The assessments of CR or PR required confirmation using bone scans.
Time Frame: Up to 46 months
Population: HER2-Positive Population. Only those participants with CR or PR were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 16 | 31
Participants
  Week 12 | 11 | 23
  Week 16 | 1 | 3
  Week 24 or longer | 4 | 5

12. Secondary Outcome: Duration of Response for the Participants With CR or PR in the HER2-Positive Population as Assessed by the Investigator
Description: Duration of response is defined as the time from the first documented evidence of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the baseline sum LD) until the first documented sign of disease progression or death due to any cause. The assessments of CR or PR required confirmation using bone scans.
Time Frame: Up to 46 months
Population: HER2-Positive Population. Only those participants with CR or PR were assessed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 16 | 31
weeks | 84.4 [29.1 to NA] — NA: Not estimable due to insufficient number of participants with events | 47.4 [25.1 to 108.0]

13. Secondary Outcome: Number of Participants With Evidence of Brain Metastases in the HER2-Positive Population
Description: The confirmation criteria for the evidence of brain metastases was the incidence of lesions occurring within any part of the central nervous system (CNS) as evidenced by radiological scans. Metastases are defined as the spread of cancer from one part of the body to another.
Time Frame: Up to 46 months
Population: HER2-Positive Population
Measure: Number; unit: participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
participants | 2 | 1

14. Secondary Outcome: Time to Progression (TTP) for the HER2-Positive Population as Assessed by the Investigator
Description: TTP is defined as the interval between the date of randomization and the earliest date of disease progression or death due to breast cancer. Disease progression was based on the assessments by the Investigator.
Time Frame: Up to 46 months
Population: HER2-Positive Population. Only those participants who experienced disease progression or died due to breast cancer were assessed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 89 | 87
weeks | 13.0 [12.0 to 23.7] | 35.4 [24.1 to 39.4]

15. Secondary Outcome: Overall Survival in the ITT Population
Description: Overall survival was defined as the time from randomization until death due to any cause.
Time Frame: From date of randomization until date of death due to any cause, assessed up to 46 months
Population: ITT Population. Only those participants who died during the study due to any cause were assessed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 234 | 240
weeks | 176.3 [156.1 to 189.7] | 170.9 [157.7 to 196.3]

16. Secondary Outcome: Overall Tumor Response (OR) for Participants With Measurable and Non-measurable Disease, Including Bone Scans, in the ITT Population as Assessed by the Investigator
Description: as for outcome 6
Time Frame: Up to 46 months
Population: ITT Population. Only those participants who achieved either a confirmed CR or PR were assessed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
percentage of participants | 27.8 | 30.5

17. Secondary Outcome: Number of Participants With Overall Tumor Response (OR) by Stratification Factors With Measurable Disease, Including Bone Scans, in the ITT Population as Assessed by the Investigator
Description: Participants were stratified based on site of disease at screening (SDS) (soft tissue or visceral or bone-only disease) and prior adjuvant endocrine therapy (PAET) (discontinuation interval [DI] =>6 months or DI <6 months). OR is defined as the number of participants achieving either a confirmed CR or PR. Response was assessed via RECIST. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the baseline sum LD. DI is defined as the time period from stopping the PEAT and the randomization date.
Time Frame: Up to 46 months
Population: ITT Population. Only those participants with some measurable disease were assessed. Response with bone scan confirmation was required. Participants with bone-only disease were excluded from the analysis because bone-only disease is non-measurable only per RECIST 1.0.
Measure: Number; unit: participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 486 | 480
participants
  SDS, Soft tissue or visceral | 170 | 190
  PAET, DI =>6 months: number analyzed (Participants) | 376 | 381
  PAET, DI =>6 months | 151 | 168
  PAET, DI <6 months: number analyzed (Participants) | 110 | 99
  PAET, DI <6 months | 19 | 22

18. Secondary Outcome: Clinical Benefit (CB) in the ITT Population as Assessed by the Investigator
Description: as for outcome 8
Time Frame: Up to 46 months
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
percentage of participants | 50.6 | 55.8

19. Secondary Outcome: Number of Participants With the Indicated Time to Response for CR or PR in the ITT Population as Assessed by the Investigator
Description: as for outcome 11
Time Frame: Up to 46 months
Population: ITT Population. Only those participants with CR or PR were assessed.
Measure: Number; unit: participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 179 | 196
participants
  Week 12 | 76 | 94
  Week 16 | 21 | 18
  Week 24 | 28 | 28
  Week 28 | 17 | 14
  Week 36 or longer | 37 | 42

20. Secondary Outcome: Duration of Response for the Participants With CR or PR in the ITT Population as Assessed by the Investigator
Description: as for outcome 12
Time Frame: Up to 46 months
Population: ITT Population. Only those participants with CR or PR response were assessed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 179 | 196
weeks | 72.6 [39.1 to 145.7] | 60.1 [36.0 to 138.9]

21. Secondary Outcome: Number of Participants With Evidence of Brain Metastases From the ITT Population
Description: as for outcome 13
Time Frame: Up to 46 months
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
participants | 4 | 6

22. Secondary Outcome: TTP for Participants From the ITT Population as Assessed by the Investigator
Description: as for outcome 14
Time Frame: Up to 46 months
Population: ITT Population. Only those participants who experienced disease progression or died due to breast cancer were assessed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 469 | 409
weeks | 47.0 [36.9 to 50.9] | 51.7 [47.6 to 59.6]

23. Secondary Outcome: Number of Participants Completing the Functional Assessment of Cancer Therapy-breast (FACT-B) Questionnaire at the Scheduled Visits
Description: Quality of Life (QOL) was assessed using the FACT-B questionnaire, which was a 37-item (27 general and 10 breast cancer-specific questions) self-reporting instrument consisting of 5 dimensions: physical-, social/family-, emotional-, functional-well being, and a breast cancer subscale. Higher scores on the FACT-B scales (each ranging from 0 [not at all] to 4 [very much]) indicate a higher QOL. The score is transformed for FACT-B and results in a total score ranging from 0 to 144. Complete: completing at least 1 question from FACT-B.
Time Frame: Day 1 (baseline) visit; Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192 visits; conclusion/withdrawal visit
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants
  Day 1, baseline | 605 | 605
  Week 12 | 460 | 476
  Week 24 | 350 | 382
  Week 36 | 291 | 294
  Week 48 | 254 | 243
  Week 60 | 199 | 183
  Week 72 | 181 | 153
  Week 84 | 144 | 119
  Week 96 | 117 | 98
  Week 108 | 80 | 62
  Week 120 | 59 | 56
  Week 132 | 43 | 43
  Week 144 | 33 | 33
  Week 156 | 22 | 21
  Week 168 | 15 | 11
  Week 180 | 11 | 5
  Week 192 | 6 | 1
  Conclusion/withdrawal | 327 | 359

24. Secondary Outcome: Adjusted Mean Change From Baseline for the FACT-B Total Score Using Observed Data
Description: Quality of Life (QOL) was assessed using the FACT-B questionnaire, which is a 37-item (27 general and 10 breast cancer-specific questions) self-reporting instrument consisting of 5 dimensions: physical-, social/family-, emotional-, functional-well being, and a breast cancer subscale. Higher scores on the FACT-B scales indicate a higher QOL; each ranging from 0 (not at all) to 4 (very much). The score is transformed for FACT-B and results in a total score ranging from 0 to 144. The FACT-B is designed to measure multidimensional QOL in participants with breast cancer.
Time Frame: Week 12, 24, 36, and 48 visits; conclusion/withdrawal visit
Population: HER2-Positive Population. Only those participants whose item response rate was greater than 80% were assessed.
Measure: Number; unit: Adjusted mean change
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 61 | 78
Adjusted mean change
  Week 12: number analyzed (Participants) | 57 | 78
  Week 12 | 1.5 | 3.3
  Week 24: number analyzed (Participants) | 36 | 53
  Week 24 | 3.8 | 1.9
  Week 36: number analyzed (Participants) | 23 | 31
  Week 36 | 3.3 | 1.4
  Week 48: number analyzed (Participants) | 22 | 23
  Week 48 | 2.9 | 0.3
  Conclusion/WD: number analyzed (Participants) | 61 | 69
  Conclusion/WD | -9.4 | -9.0

25. Secondary Outcome: Adjusted Mean Change From Baseline for the Functional Assessment of Cancer Therapy-General (FACT-G) Score Using Observed Data
Description: FACT-G is a subscale of the FACT-B QOL questionnaire and consists of 27 questions grouped into 4 domains that measure a participant's physical, functional, social and family, and emotional well-being. FACT-G is assessed on a five-point Likert-type scale, with scores ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The total score is calculated as the sum of the item scores on the subscale; the total ranges from 0 to 108, with higher score indicating a better quality of life.
Time Frame: Week 12, 24, 36, and 48 visits; conclusion/withdrawal visit
Population: HER2-Positive Population. Only those participants whose item response rate was greater than 80% were assessed.
Measure: Number; unit: Adjusted mean change
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 63 | 79
Adjusted mean change
  Week 12: number analyzed (Participants) | 60 | 79
  Week 12 | 1.6 | 1.5
  Week 24: number analyzed (Participants) | 37 | 54
  Week 24 | 2.2 | 0.6
  Week 36: number analyzed (Participants) | 24 | 33
  Week 36 | 2.6 | 0.9
  Week 48: number analyzed (Participants) | 23 | 25
  Week 48 | 2.0 | -0.9
  Conclusion/WD: number analyzed (Participants) | 63 | 71
  Conclusion/WD | -7.8 | -8.5

26. Secondary Outcome: Adjusted Mean Change From Baseline for the Trial Outcome Index (TOI) Score Using Observed Data
Description: The TOI score is the sum of the physical well-being, functional well-being, and breast cancer unweighted subscale scores. The total TOI score ranges from 0 to 92, with higher scores representing a better quality of life.
Time Frame: Week 12, 24, 36, and 48 visits; conclusion/withdrawal visit
Population: HER2-Positive Population. Only those participants whose item response rate was greater than 80% were assessed.
Measure: Number; unit: Adjusted mean change
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 62 | 77
Adjusted mean change
  Week 12: number analyzed (Participants) | 59 | 77
  Week 12 | -0.3 | 2.7
  Week 24: number analyzed (Participants) | 37 | 52
  Week 24 | 3.9 | 2.0
  Week 36: number analyzed (Participants) | 24 | 28
  Week 36 | 3.3 | 0.8
  Week 48: number analyzed (Participants) | 22 | 23
  Week 48 | 2.2 | -0.7
  Conclusion/WD: number analyzed (Participants) | 62 | 67
  Conclusion/WD | -6.2 | -6.4

27. Secondary Outcome: Number of Participants Classified as QOL Responders Based on the FACT-B, FACT-G, and TOI Total Scores
Description: A minimally important difference (MID) is the smallest difference in a score for a measure of QOL that corresponds to a difference in function or clinical course. Responders are defined as participants with an MID => 8 for the FACT-B score, and an MID =>6 for the FACT-G and TOI scores.
Time Frame: Up to 46 months
Population: HER2-Positive Population. Only those participants with a baseline score and at least one post-baseline score were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 87 | 99
Participants
  FACT-B total, =>8 (MID upper bound): number analyzed (Participants) | 85 | 98
  FACT-B total, =>8 (MID upper bound) | 29 | 33
  FACT-G, =>6 (MID upper bound) | 29 | 38
  TOI, =>6 (MID upper bound): number analyzed (Participants) | 87 | 97
  TOI, =>6 (MID upper bound) | 29 | 33

28. Secondary Outcome: Number of Participants With Clinical Benefit Categorized by HER2 Fluorescence in Situ Hybridization (FISH) Status
Description: Clinical benefit: participants with CR, PR, or SD for =>6-month period. FISH testing measures the amount of the HER2 gene in each cell. This gene is responsible for the overproduction of the HER2 protein. FISH-positive: excessive amounts of the gene are present; FISH-negative: normal levels of the gene are present.
Time Frame: Up to 46 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants
  FISH status, Positive: number analyzed (Participants) | 96 | 97
  FISH status, Positive | 28 | 49
  FISH status, Negative: number analyzed (Participants) | 412 | 422
  FISH status, Negative | 237 | 245
  FISH status, missing: number analyzed (Participants) | 136 | 123
  FISH status, missing | 61 | 64

29. Secondary Outcome: Number of Participants With Clinical Benefit Categorized by HER2 ImmunoHistoChemistry (IHC) Intensity
Description: IHC is a commonly used test to assess the amount of the HER2 receptor protein on the surface of the cancer cells. The IHC test results in a score of 0 to 3+, which indicates the amount of HER2 receptor protein on the cells in a sample of breast cancer tissue. Tissue scores of 0 to 1+ indicate HER2 negativity; scores of 2+ and 3+ indicate HER2 positivity. Clinical benefit is defined as participants with CR, PR, or SD for =>6-month period.
Time Frame: Up to 46 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants
  IHC Intensity 0: number analyzed (Participants) | 153 | 177
  IHC Intensity 0 | 74 | 106
  IHC Intensity 1: number analyzed (Participants) | 189 | 190
  IHC Intensity 1 | 108 | 106
  IHC Intensity 2: number analyzed (Participants) | 165 | 146
  IHC Intensity 2 | 94 | 85
  IHC Intensity 3: number analyzed (Participants) | 64 | 61
  IHC Intensity 3 | 16 | 26
  IHC Intensity Missing: number analyzed (Participants) | 73 | 68
  IHC Intensity Missing | 34 | 35

30. Secondary Outcome: Number of Participants With Response in Participants With Baseline Serum HER2 Extracellular Domain (ECD) Baseline Values Greater Than 15 Nanograms Per Milliliter (ng/mL) and 15 ng/mL or Lower
Description: The HER2 ECD is a glycoprotein that can be shed from the cell surface into the blood of normal individuals and can be elevated in different pathologic conditions. The serum HER2 ECD level generally reflects the tissue HER2 status. The HER2 ECD is quantified in serum with an enzyme-linked immunosorbent assay (ELISA). Non-Evaluable (NE): any participant who could not be classified as CR, PR, SD, or PD.
Time Frame: Up to 46 months
Population: HER2-Positive Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 108 | 111
Participants
  >15 ng/mL, CR/PR: number analyzed (Participants) | 53 | 34
  >15 ng/mL, CR/PR | 3 | 9
  >15 ng/mL, SD: number analyzed (Participants) | 53 | 34
  >15 ng/mL, SD | 11 | 13
  >15 ng/mL, PD/NE: number analyzed (Participants) | 53 | 34
  >15 ng/mL, PD/NE | 39 | 12
  =<15 ng/mL, CR/PR: number analyzed (Participants) | 51 | 70
  =<15 ng/mL, CR/PR | 12 | 17
  =<15 ng/mL, SD: number analyzed (Participants) | 51 | 70
  =<15 ng/mL, SD | 23 | 30
  =<15 ng/mL, PD/NE: number analyzed (Participants) | 51 | 70
  =<15 ng/mL, PD/NE | 16 | 23

31. Secondary Outcome: Number of HER2-Negative Participants at Baseline With and Without Seroconversion to a Status of HER2 Positive
Description: Participants who had a HER2-negative tumor status based on baseline tissue with baseline serum HER2 ECD values =<15 ng/mL but later had at least two consecutive serum HER2 ECD values >15 ng/mL experienced seroconversion.
Time Frame: Up to 46 months
Population: HER2-Negative Population: all randomized participants regardless of whether or not study treatment had been received and who at baseline were evaluated by the central laboratory to have retrospectively documented non-amplification or missing amplification of HER2 by FISH (<2.0) and documented IHC scores of 0, 1+, 2+, or missing in tumor tissue.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 474 | 478
Participants
  Seroconversion, No | 323 | 140
  Seroconversion, Yes | 52 | 219
  Missing | 99 | 119

32. Secondary Outcome: Time to Seroconversion for Participants Who Were HER2 Negative at Baseline But Became HER2 Positive
Description: Time to seroconversion was defined as the time from the date of randomization until the first instance of serum HER2 (>15 ng/mL) on two consecutive occasions.
Time Frame: Up to 46 months
Population: HER2-Negative Population. Only those participants who had a HER2-negative tumor status based on baseline tissue with baseline serum HER2 ECD values =<15 ng/mL but later had at least two consecutive serum HER2 ECD values >15 ng/mL were assessed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 52 | 219
Weeks | NA [NA to NA] — As >80% of the participants were censored, no median or confidence intervals could be established. | 36.1 [24.0 to 48.9]

33. Secondary Outcome: Number of Participants With the Indicated Expression of Tumor by Epidermal Growth Factor Receptor (ErbB1/HER1/EGFR) at Baseline
Description: EGFR is a cell surface receptor tyrosine kinase expressed in certain types of tumors. Depending upon the staining intensity, EGFR was graded as follows: 0=absence of membrane staining above background in all tumor cells; EGFR-positive=staining is defined as any IHC staining of tumor cell membranes above background level, whether it is complete or incomplete circumferential staining (1+, 2+, 3+).
Time Frame: Baseline
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 644 | 642
Participants
  EGFR, 0: number analyzed (Participants) | 576 | 580
  EGFR, 0 | 513 | 522
  EGFR, 1+: number analyzed (Participants) | 576 | 580
  EGFR, 1+ | 43 | 45
  EGFR, 2+: number analyzed (Participants) | 576 | 580
  EGFR, 2+ | 17 | 12
  EGFR, 3+: number analyzed (Participants) | 576 | 580
  EGFR, 3+ | 3 | 1

34. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 663.9 weeks (treatment duration ranged from 0.1 to 659.9 weeks).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 14 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 663 weeks (on-treatment), up to approximately 14 years (study duration)
Population: Clinical database population; all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
Number analyzed (Participants) | 624 | 654
Participants
  On-treatment deaths | 23 | 18
  All deaths | 484 | 488

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of 663.9 weeks (treatment duration ranged from 0.1 to 659.9 weeks).
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up. Maximum exposure to Lapatinib = 612 weeks (Lapatinib + Letrozole treatment group). Maximum exposure to Letrozole = 659.7 weeks (Placebo + Letrozole treatment group) and 612 weeks (Lapatinib + Letrozole treatment group).
Arm/Group | Placebo + Letrozole 2.5 mg | Lapatinib 1500 mg + Letrozole 2.5 mg
All-Cause Mortality (participants affected / at risk) | 23/624 | 18/654
Serious Adverse Events (participants affected / at risk) | 103/624 | 150/654
Other Adverse Events (participants affected / at risk) | 481/624 | 589/654
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Letrozole 2.5 mg (N=624) | Lapatinib 1500 mg + Letrozole 2.5 mg (N=654)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Jaundice (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Dyspnoea (Cardiac disorders) | 5 | 6
Left ventricular dysfunction (Cardiac disorders) | 1 | 7
Left ventricular failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Peripheral swelling (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 3 | 1
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0
Carcinoid tumour (Endocrine disorders) | 0 | 1
Hypercalcaemia (Endocrine disorders) | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Eye injury (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 3
Clostridium difficile colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colon cancer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 15
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 5
Oral infection (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Peritonitis bacterial (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 9
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 3 | 4
Complication associated with device (General disorders) | 1 | 0
Decreased appetite (General disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 4
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1
Gallbladder pain (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Crohn's disease (Immune system disorders) | 1 | 0
Dermatomyositis (Immune system disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 4
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 4 | 3
Pyelonephritis (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 6
Urosepsis (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Accidental poisoning (Injury, poisoning and procedural complications) | 1 | 0
Catheter site infection (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatotoxicity (Injury, poisoning and procedural complications) | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural infection (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0
Toxic skin eruption (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 1
Wound infection (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 8 | 17
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency anaemia (Metabolism and nutrition disorders) | 0 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Humerus fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Confusional state (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Meningioma (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Device breakage (Product Issues) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hepatorenal failure (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Hypercreatininaemia (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Pelvic pain (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Breast abscess (Reproductive system and breast disorders) | 0 | 1
Breast cellulitis (Reproductive system and breast disorders) | 1 | 1
Ovarian enlargement (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 0 | 1
Incision site cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Infected skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Malignant melanoma (Skin and subcutaneous tissue disorders) | 0 | 1
Paronychia (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Acute myocardial infarction (Vascular disorders) | 1 | 0
Angina unstable (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Gastrointestinal haemorrhage (Vascular disorders) | 1 | 2
Haematemesis (Vascular disorders) | 0 | 2
Haematochezia (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemoptysis (Vascular disorders) | 0 | 2
Haemorrhoids thrombosed (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 2 | 0
Melaena (Vascular disorders) | 0 | 1
Myocardial infarction (Vascular disorders) | 1 | 1
Pulmonary hypertension (Vascular disorders) | 0 | 1
Rectal haemorrhage (Vascular disorders) | 0 | 2
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Uterine haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Letrozole 2.5 mg (N=624) | Lapatinib 1500 mg + Letrozole 2.5 mg (N=654)
Anaemia (Blood and lymphatic system disorders) | 28 | 52
Dyspnoea (Cardiac disorders) | 68 | 58
Abdominal pain (Gastrointestinal disorders) | 28 | 48
Abdominal pain upper (Gastrointestinal disorders) | 16 | 36
Constipation (Gastrointestinal disorders) | 64 | 45
Diarrhoea (Gastrointestinal disorders) | 109 | 393
Dyspepsia (Gastrointestinal disorders) | 28 | 56
Nausea (Gastrointestinal disorders) | 123 | 190
Stomatitis (Gastrointestinal disorders) | 8 | 34
Vomiting (Gastrointestinal disorders) | 69 | 101
Asthenia (General disorders) | 62 | 76
Decreased appetite (General disorders) | 55 | 80
Fatigue (General disorders) | 98 | 124
Mucosal inflammation (General disorders) | 11 | 37
Pyrexia (General disorders) | 32 | 42
Nasopharyngitis (Infections and infestations) | 44 | 50
Upper respiratory tract infection (Infections and infestations) | 32 | 31
Urinary tract infection (Infections and infestations) | 44 | 35
Alanine aminotransferase increased (Investigations) | 28 | 58
Aspartate aminotransferase increased (Investigations) | 24 | 54
Blood alkaline phosphatase increased (Investigations) | 15 | 34
Weight decreased (Investigations) | 13 | 35
Oedema peripheral (Metabolism and nutrition disorders) | 46 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 135 | 112
Back pain (Musculoskeletal and connective tissue disorders) | 91 | 99
Bone pain (Musculoskeletal and connective tissue disorders) | 48 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 33
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 34 | 30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 49 | 52
Myalgia (Musculoskeletal and connective tissue disorders) | 41 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 65 | 67
Dizziness (Nervous system disorders) | 46 | 44
Headache (Nervous system disorders) | 79 | 84
Insomnia (Nervous system disorders) | 50 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 89 | 71
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 61
Acne (Skin and subcutaneous tissue disorders) | 4 | 39
Alopecia (Skin and subcutaneous tissue disorders) | 39 | 74
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 82
Erythema (Skin and subcutaneous tissue disorders) | 9 | 33
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 63
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 50 | 76
Rash (Skin and subcutaneous tissue disorders) | 56 | 223
Hot flush (Vascular disorders) | 80 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.